CLINICAL TRIAL: NCT04800133
Title: To Compare the Reactogenicity and Immunogenicity of Recommended COVID-19 Vaccines in Young Adolescents and Children in Hong Kong
Brief Title: Covid-19 Vaccination in Adolescents and Children
Acronym: COVAC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COVAC01
Record Dates: First submitted 2021-03-01; First posted 2021-03-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; sinovac COVID-19 vaccine; Injections, Intradermal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- BNT162b2 (adult/adolescent) (Experimental): BNT162b2, tozinameran by Fosun/BioNTech Intramuscular injection (or intradermal for immunocompromised patients; or by graded challenge with history of non-severe allergy to PEG-containing drugs) 30ug/0.3ml per dose 3 doses, or 4 for immunocompromised patients; or 1/2 dose for patients with prior COVID-19
  Interventions: Biological: Tozinameran
- CoronaVac (intramuscular) (Experimental): CoronaVac by SinoVac Intramuscular injection 3ug/0.5ml per dose 3 doses, or 4 for immunocompromised patients; or 1/2 dose for patients with prior COVID-19
  Interventions: Biological: CoronaVac
- CoronaVac (intradermal) (Experimental): CoronaVac by SinoVac Intradermal injection 3ug/0.5ml per dose 3 doses, or 4 for immunocompromised patients; or 1/2 dose for patients with prior COVID-19
  Interventions: Biological: CoronaVac, intradermal
- BNT162b2 (paediatric) (Experimental): BNT162b2, tozinameran by Fosun/BioNTech Intramuscular injection (for immunocompromised patients only) 10ug/0.1ml per dose 4 doses for immunocompromised patients
  Interventions: Biological: Tozinameran

INTERVENTIONS:
Biological: Tozinameran — mRNA vaccine developed by BioNTech against COVID-19
  Other Names: BNT162b2
  Arms: BNT162b2 (adult/adolescent); BNT162b2 (paediatric)
Biological: CoronaVac — Inactivated virus vaccine developed by SinoVac against COVID-19, intramuscular
  Arms: CoronaVac (intramuscular)
Biological: CoronaVac, intradermal — Inactivated virus vaccine developed by SinoVac against COVID-19, intradermal
  Arms: CoronaVac (intradermal)

SUMMARY:
Objectives To assess the reactogenicity, measure the adaptive immune responses and track the long-term immune memory in healthy children and adults as well as pediatric patients receiving the COVID-19 vaccines-BNT162b2, CoronaVac-chosen by the Hong Kong Government; to compare the reactogenicity and immunogenicity across the vaccines used for these children and adults.

Hypothesis to be tested The safety profile and the magnitude and durability of immune responses to the COVID-19 vaccines in children are non-inferior to those in adults.

Design and subjects A single-site, comparative nonrandomised clinical trial for 450 healthy individuals or patients under 18 years old and one or both healthy parents and unrelated adults to receive one of COVID-19 vaccines by intramuscular injection (and intradermal injection)

Instruments Mobile app for subjects to record adverse effects, enzyme-linked immunosorbent assay, plaque reduction neutralization assay, luciferase immunoprecipitation system assay and flow cytometry.

Interventions BNT162b2 and CoronaVac, by intramuscular or intradermal route

Main outcome measures Types and frequencies of adverse effects within 7 days, and changes and peaks of antibody levels and antigen-specific memory T cell responses for 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. informed consent from the parents or a legally acceptable representative for an underage participant
2. biological parents of students enrolled in the trial or unrelated healthy adults
3. ability to adhere to the follow-up schedules
4. willingness to report reactogenicity daily for 7 days post dose 1, 2 and 3 (and 4) proactively
5. willingness to receive that vaccine available for that particular recruitment period (as student-parent pair, if applicable)
6. good past health, including pre-existing clinically stable disease, such as paediatric or immune disorders
7. prior COVID-19 (for COVID-19 survivor subgroup)

Exclusion Criteria:

1. reported pregnancy or breastfeeding

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1018 (Actual)
Dates: Start 2021-05-08 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse reactions | 7 days post-doses 1, 2 and 3 (and 4)
  Percentage of occurrence, types, duration and severity of adverse reactions occurring within 7 days
Binding antibody response | 1 month post-dose 1, and 1, 6, 18, and 36 months post-dose 3 (and 2 weeks after dose 4)
  Geometric mean levels of SARS-CoV2 S and S-RBD-specific binding antibody and related markers as determined by Enzyme-linked Immunosorbent Assay
Neutralizing antibody response | 1 month post-dose 1, and 1, 6, 18, and 36 months post-dose 3 (and 2 weeks after dose 4)
  Geometric mean levels and geometric mean fold rise of SARS-CoV2 neutralizing antibodies as determined by plaque reduction neutralization assay and surrogate assays
T cell response | 1 month post-dose 1, and 1, 6, 18, and 36 months post-dose 3 (and 2 weeks after dose 4)
  Geometric mean percentage of CD4 and CD8 T cells specific to SARS-CoV2 S (and N and M) protein

SECONDARY OUTCOMES:
Vaccine breakthrough | Throughout the study period, until 36 months post-dose 3/4
  Incidence of COVID-19 in participants throughout study period as self-reported or as determined by Luciferase Immunoprecipitation Systems assay/ELISA
Adverse events | Throughout the study period, until 36 months post-dose 3/4
  Percentage of occurrence, types, duration and severity of adverse events and severe adverse events throughout study period
Binding anti-N antibody response | 1 month post-dose 1, and 1, 6, 18, and 36 months post-dose 3 (and 2 weeks after dose 4)
  Geometric mean levels and geometric mean fold rise of SARS-CoV2 N-specific binding antibody as determined by Enzyme-linked Immunosorbent Assay in Arm C participants receiving CoronaVac

CONTACTS AND LOCATIONS:
Overall Officials: Yu Lung Lau, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosa Duque JS, Wang X, Leung D, Cheng SMS, Cohen CA, Mu X, Hachim A, Zhang Y, Chan SM, Chaothai S, Kwan KKH, Chan KCK, Li JKC, Luk LLH, Tsang LCH, Wong WHS, Cheang CH, Hung TK, Lam JHY, Chua GT, Tso WWY, Ip P, Mori M, Kavian N, Leung WH, Valkenburg S, Peiris M, Tu W, Lau YL. Immunogenicity and reactogenicity of SARS-CoV-2 vaccines BNT162b2 and CoronaVac in healthy adolescents. Nat Commun. 2022 Jun 28;13(1):3700. doi: 10.1038/s41467-022-31485-z. PMID 35764637